CLINICAL TRIAL: NCT01365585
Title: Evaluate The Clinical Effectiveness, Safety And Tolerability Of Sildenafil Used In Doses ≥20mg TID For The Treatment Of Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481297
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; sildenafil citrate; Revatio
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sildenafil ≥20mg three times daily: Subjects receiving sildenafil ≥20mg three times daily for the treatment of PAH
  Interventions: Drug: sildenafil citrate

INTERVENTIONS:
Drug: sildenafil citrate — Sildenafil citrate, 20mg oral tablets, taken at least three times daily

SUMMARY:
The objective of this observational study is to gain clinical insight on the actual use of sildenafil citrate (Revatio™) for the treatment of pulmonary arterial hypertension (PAH). The primary objective is to assess effectiveness and safety of sildenafil at doses ≥20mg three times daily for the treatment of PAH.

DETAILED DESCRIPTION:
The study design proposed is a retrospective chart review going back five years (01 April 2006 estimate) from the time of study initiation (31 March 2011 estimate). Within this five-year period, study index will occur the first time an adult patient begins sildenafil for the treatment of PAH for a period of at least three months. The patient has to be taking sildenafil at doses ≥ 20mg tid for the treatment of PAH.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age at study index;
* Patients must have a diagnosis of PAH. PAH is conventionally defined as a mean pulmonary arterial pressure (PAP) of > 25 mmHg and a pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg and a pulmonary vascular resistance (PVR) ≥ 240 dynes/s/cm-5 at right heart catheterization;
* Patients must have initiated sildenafil for the treatment of their PAH; at dose ≥ 20 mg tid within 5 years prior to study initiation

Exclusion Criteria:

* Patient has known contraindications to sildenafil at study index;
* Patient participated in an investigational study of sildenafil treatment for PAH during the period beginning 6 months prior to study index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 18 years of age diagnosed with pulmonary arterial hypertension (PAH; per Dana Point classification) and treated with sildenafil citrate for their PAH
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Medizinische Hochschule Hannover, Hanover, Germany
- Mater Misericordiae Hospital, Dublin, Ireland

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil: Participants who received sildenafil greater than or equal to 20 milligram (mg) three times daily as per Summary of Product Characteristics (SmPC) for the treatment of pulmonary arterial hypertension (PAH) for a period of at least 3 months, were observed retrospectively for 5 years.
Period: Overall Study
Arm/Group | Sildenafil
Started | 227
Completed | 227
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sildenafil
Number analyzed (Participants) | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (14.37)
Sex/Gender, Customized [Number; unit: participants] — For baseline characteristic gender, number of participants evaluable was 226.
  participants
    Female | 145
    Male | 81
Six-Minute Walk Distance (6MWD) [Mean (Standard Deviation); unit: meter] — 6MWD was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. Number of participants evaluable for this measure was 176.
  meter | 331.7 (117.42)
New York Heart Association, World Health Organization (NYHA/WHO) Functional Class [Number; unit: participants] — NYHA/WHO functional classification for PAH range from Class I (no limitation in physical activity, no dyspnea with normal activity) to Class IV (can not perform a physical activity without any symptoms, dyspnea at rest). Number of participants in each functional class was reported. Number of participants evaluable for this measure was 216.
  participants
    Class I | 1
    Class II | 39
    Class III | 163
    Class IV | 13
Right Atrial Pressure (RAP) [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] — RAP was measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position. Number of participants evaluable for this measure was 50.
  millimeters of mercury (mmHg) | 6.6 (4.85)
Mean Pulmonary Arterial Pressure (mPAP) at rest [Mean (Standard Deviation); unit: mmHg] — mPAP was measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position. Number of participants evaluable for this measure was 56.
  mmHg | 44.8 (12.37)
Pulmonary Vascular Resistance (PVR) [Mean (Standard Deviation); unit: dynes*second/centimeter^5] — PVR: calculated by subtracting PCWP from mPAP and dividing by cardiac output in pulmonary circulation (COpulm). Number of participants evaluable for this measure was 48.
  dynes*second/centimeter^5 | 612.8 (250.54)
Cardiac Index (CI) [Mean (Standard Deviation); unit: (Liter/minute)/square meter([L/min]/m^2)] — CI: calculated as cardiac output in systemic circulation (COsys) divided by body surface area (BSA). Number of participants evaluable for this measure was 44.
  (Liter/minute)/square meter([L/min]/m^2) | 2.5 (1.51)
Pulmonary Capillary Wedge Pressure (PCWP) [Mean (Standard Deviation); unit: mmHg] — PCWP was measured by pulmonary artery catheterization and provided an indirect measure of left atrial pressure. Number of participants evaluable for this measure was 44.
  mmHg | 7.6 (3.84)
Borg Dyspnea Index [Mean (Standard Deviation); unit: units on a scale] — Borg dyspnea scale: 10-point scale where following scores stands for severity of dyspnea: 0=no breathlessness at all; 0.5=very very slight (just noticeable); 1=very slight; 2=slight breathlessness; 3=moderate; 4=some what severe; 5=severe; 7=very severe breathlessness; 9=very very severe (almost maximum) and 10=maximum. Participants evaluable=158.
  units on a scale | 3.7 (1.91)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD) at Year 1
Description: 6MWD was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed.
Time Frame: Baseline, Year 1
Population: Analysis population included all participants who satisfied the eligibility criteria for the study. Here, 'N' (number of participants analyzed) included those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Sildenafil
Number analyzed (Participants) | 132
meter | 29.4 (81.38)

2. Primary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD) at Year 2
Description: as for outcome 1
Time Frame: Baseline, Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Sildenafil
Number analyzed (Participants) | 74
meter | 20.8 (83.82)

3. Primary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD) at Year 3
Description: as for outcome 1
Time Frame: Baseline, Year 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Sildenafil
Number analyzed (Participants) | 31
meter | 8.7 (73.82)

4. Primary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD) at Year 4
Description: as for outcome 1
Time Frame: Baseline, Year 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Sildenafil
Number analyzed (Participants) | 9
meter | -50.2 (86.24)

5. Secondary Outcome: Change From Baseline in New York Heart Association, World Health Organization (NYHA/WHO) Functional Class in Participants With Pulmonary Arterial Hypertension (PAH) at Year 1, 2, 3 and 4
Description: NYHA/WHO functional classification for PAH range from Class I (no limitation in physical activity, no dyspnea with normal activity) to Class IV (can not perform a physical activity without any symptoms, dyspnea at rest). Improvement=reduction in functional class, deterioration = increase in functional class, no change = no change in functional class. Number of participants in each functional class was reported.
Time Frame: Baseline, Year 1, 2, 3, 4
Population: Analysis population included all participants who satisfied the eligibility criteria for the study. Here, 'N' (number of participants analyzed) included those participants who were evaluable for this measure. Here, 'n' included those participants who were evaluable for this measure at specified time points.
Measure: Number; unit: participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 214
participants
  Year 1: Improved >1 class (n=214) | 3
  Year 1: Improved 1 class (n=214) | 36
  Year 1: No change (n=214) | 140
  Year 1: Worsened 1 class (n=214) | 12
  Year 1: Worsened >1 class (n=214) | 5
  Year 2: Improved >1 class (n=156) | 1
  Year 2: Improved 1 class (n=156) | 27
  Year 2: No change (n=156) | 100
  Year 2: Worsened 1 class (n=156) | 7
  Year 2: Worsened >1 class (n=156) | 4
  Year 3: Improved >1 class (n=88) | 1
  Year 3: Improved 1 class (n=88) | 12
  Year 3: No change (n=88) | 57
  Year 3: Worsened 1 class (n=88) | 7
  Year 3: Worsened >1 class (n=88) | 0
  Year 4: Improved >1 class (n=45) | 0
  Year 4: Improved 1 class (n=45) | 6
  Year 4: No change (n=45) | 27
  Year 4: Worsened 1 class (n=45) | 2
  Year 4: Worsened >1 class (n=45) | 0

6. Secondary Outcome: Change From Baseline in Right Atrial Pressure (RAP) at Year 1, 2, 3 and 4
Description: RAP was measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position.
Time Frame: Baseline, Year 1, 2, 3, 4
Population: Data was not summarized because results were available for very few participants and were insufficient for analysis.
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Mean Pulmonary Arterial Pressure (mPAP) at Rest at Year 1, 2, 3 and 4
Description: mPAP was measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position.
Time Frame: Baseline, Year 1, 2, 3, 4
Population: Data was not summarized because results were available for very few participants and were insufficient for analysis.
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) at Year 1, 2, 3 and 4
Description: PVR: calculated by subtracting PCWP from mPAP and dividing by cardiac output in pulmonary circulation (COpulm).
Time Frame: Baseline, Year 1, 2, 3, 4
Population: Data was not summarized because results were available for very few participants and were insufficient for analysis.
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in Cardiac Index (CI) at Year 1, 2, 3 and 4
Description: CI: calculated as COsys divided by BSA.
Time Frame: Baseline, Year 1, 2, 3, 4
Population: Data was not summarized because results were available for very few participants and were insufficient for analysis.
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Pulmonary Capillary Wedge Pressure (PCWP) at Year 1, 2, 3 and 4
Description: PCWP was measured by pulmonary artery catheterization and provided an indirect measure of left atrial pressure.
Time Frame: Baseline, Year 1, 2, 3, 4
Population: Data was not summarized because results were available for very few participants and were insufficient for analysis.
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline in Borg Dyspnea Index at Year 1, 2, 3 and 4
Description: Borg dyspnea scale: 10-point scale where following scores stands for severity of dyspnea: 0=no breathlessness at all;0.5=very very slight (just noticeable); 1=very slight; 2=slight breathlessness; 3=moderate; 4=some what severe; 5=severe; 7=very severe breathlessness; 9=very very severe (almost maximum) and 10=maximum.
Time Frame: Baseline, Year 1, 2, 3, 4
Population: Analysis population included all participants who satisfied the eligibility criteria for the study. Here, 'N' (number of participants analyzed) included those participants who were evaluable for this measure. 'n' included those participants who were evaluable for this measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil
Number analyzed (Participants) | 118
units on a scale
  Change at Year 1 (n=118) | -0.4 (1.88)
  Change at Year 2 (n=65) | 0.0 (2.01)
  Change at Year 3 (n=27) | 0.3 (1.82)
  Change at Year 4 (n=8) | 0.4 (1.92)

ADVERSE EVENTS:
Description: Only those adverse events that were determined to be related to sildenafil by the investigator were reported in this observational retrospective study.
Arm/Group | Sildenafil
Serious Adverse Events (participants affected / at risk) | 0/227
Other Adverse Events (participants affected / at risk) | 11/227
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil (N=227)
Ankle oedema, facial flushing (General disorders) | 1
Back pain or dizziness or eyesight (General disorders) | 1
Cough (General disorders) | 1
Dizziness (General disorders) | 1
Gastro-intestinal symptoms (General disorders) | 1
Head fuzzy/mild headache/mild flushing/mild nasal congestion (General disorders) | 1
Headache, diarrhoea and anxiety (General disorders) | 1
Mild headache/increased heart rate (General disorders) | 1
Nasal stuffiness/headache (General disorders) | 1
Nose bleeds (General disorders) | 1
Rash/itch (severe) (General disorders) | 1
Red face/peripheral oedema (General disorders) | 1
Vague upper abdominal discomfort by suspected pancreatic cancer (General disorders) | 1
Worsening of PAH (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.